CLINICAL TRIAL: NCT02843945
Title: Initial Feasibility Study to Evaluate the Safety and Efficacy of the Permanently Implantable LDR CivaSheet® in Combination With External Beam Radiation in the Treatment of Pancreatic Cancer
Brief Title: Initial Feasibility Study to Treat Borderline Resectable Pancreatic Cancer With a Planar LDR Source
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CivaTech Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT004
Record Dates: First submitted 2016-06-16; First posted 2016-07-26 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer
Keywords: brachytherapy; CivaSheet; CivaTech; whipple; radiation; borderline resectable; locally advanced; Pd-103; intraoperative radiation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation Phase I followed by a feasibility trial in Phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Directional Brachytherapy Source Implant (Experimental): Patients undergoing a pancreatic cancer resection will receive a CivaSheet LDR directional brachytherapy implant at the time of surgery. The directional nature of the FDA cleared CivaSheet is expected to allow physicians to increase the radiation dose given to the surgical margin safely, reducing risk of recurrence without increasing radiation side effects.
  Interventions: Device: Directional Brachytherapy Source Implant

INTERVENTIONS:
Device: Directional Brachytherapy Source Implant — The FDA Cleared CivaSheet Directional Pd103 Brachytherapy Source is a planar radiaiton source which utilizes gold shielding in its construction. This device is radioactive on one side only, and is capable of safely delivering high doses of radiation to target areas even when placed directly adjacent to sensitive, healthy tissue or critical structures.

SUMMARY:
Initial study to evaluate local control and the preferred method of attachment of the CivaSheet in the setting of suspected close or positive margins at the time of surgical tumor removal.

DETAILED DESCRIPTION:
This is a Feasibility study to determine the safety and efficacy of a new brachytherapy device that provides unidirectional radiation which utilizes active components (Palladium-103) of standard devices in a novel configuration.This pilot study may benefit pancreatic cancer patients by reducing the radiation dose to adjacent critical structures, while giving a therapeutic dose to diseased tissue, such as at a surgical margin. The appropriate dose and local control rate will be recorded the primary endpoint in order to provide an efficacy assessment.

ELIGIBILITY:
Inclusion Criteria:

* • Subject signed inform consent

  * Age > 18 years
  * Not pregnant or breast feeding
  * Patient capable of undergoing anesthesia
  * Patient selected to undergo Whipple procedure or distal pancreatectomy
  * Patient does not have metastatic disease
  * Patients will have close margins
  * No prior radiation therapy to the region for separate cancer
  * Confirmed diagnosis of borderline resectable or locally advanced pancreatic adenocarcinoma
  * Patient Received neoadjuvant chemoradiation (4-10 weeks prior to surgery)
  * Chemotherapy was administered for 2-6 cycles with any combination of the following agents:
  * Gemcitabine + nb-paclitaxel
  * FOLFIRINOX
  * Neoadjuvant Chemoradiation was administered as IMRT or 3DCRT (up to 56 Gy), or SBRT (up to 36 Gy) with Pre-operative External beam dose (NCCN)
  * up to 56 Gy (1.8-2.0 Gy per fractions) with concurrent gemcitabine, capecitabine, or infusional 5-fluorouracil

Exclusion Criteria:

* Not surgical candidate
* Any other invasive cancer in the past 5 years, except basal cell or squamous cell skin cancer
* An IRE candidate (IRE is Percutaneous irreversible electroporation)
* Recurrent or previously resected tumors
* Documented History of Alcoholism and or drug abuse
* Participant in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety of CivaSheet Radiation Treatement | 1 Year
  Patients will be monitored for any adverse radiation toxicity effects from the CivaSheet device.

SECONDARY OUTCOMES:
Efficacy of CivaSheet Radiation Treatment | 1 Year
  Patients will be monitored for one year to determine the local cancer recurrence rate
Morbidity of patients following surgery and radiation | 2 Year
  2 year survival rates for patients post surgery and CivaSheet radiation treatment
Post Operative Radiation Dosimetry Calculation | 1 Month
  Post procedure 3D treatment planning will be performed to determine if the radiation dose delivered was satisfactory
Length of Hospital Stay | 1 Month
  Length of hospital stay will be monitored to determine if CivaSheet radiation treatment alters the typical length of hospital stay for patients after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (6):
- United States (6):
  - Tampa General Hospital, Tampa, Florida
  - Rush University Cancer Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University Medical Center LSU, New Orleans, Louisiana
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No